CLINICAL TRIAL: NCT04700046
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Investigate the Efficacy and Safety of Mexiletine During 26 Weeks of Treatment in Patients With Myotonic Dystrophy Type 1 and Type 2 [The MIND Study]
Brief Title: Study to Investigate the Efficacy and Safety of Mexiletine in Patients With Myotonic Dystrophy Type 1 and Type 2
Acronym: MIND
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Assessing novel alternative study designs and regulatory pathways
Sponsor: Lupin Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEX-DM-301
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Myotonic Dystrophy Type 1 and Type 2
MeSH Terms: conditions — Myotonic Dystrophy | interventions — Mexiletine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mexiletine (Active Comparator): Mexiletine 167 mg (equivalent to mexiletine HCl 200 mg)
  Interventions: Drug: Mexiletine 167 mg
- Placebo (Placebo Comparator): The placebo capsules contain the same ingredients as the active formulation with the exception of mexiletine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mexiletine 167 mg — Mexiletine 167 mg (equivalent to mexiletine HCl 200 mg) immediate release, oral capsules.
  Arms: Mexiletine
Drug: Placebo — The placebo capsules contain the same ingredients as the active formulation with the exception of mexiletine
  Arms: Placebo

SUMMARY:
A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Investigate the Efficacy and Safety of Mexiletine During 26 Weeks of Treatment in Patients with Myotonic Dystrophy Type 1 and Type 2 [The MIND Study]

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group, placebo-controlled study intended to evaluate the safety and efficacy of mexiletine in patients with myotonic dystrophy type 1 and type 2 (DM1 and DM2). The study will consist of a 4-week screening period and a 26-week treatment phase with patient visits as screening, baseline, weeks 1, 2, 6, 14, 18, and 26. Eligible patients will be randomized to mexiletine or placebo in a 1:1 ratio. Approximately 158 DM1 patients (79 active: 79 placebo) are planned to be enrolled across 10-15 experienced investigational centers in Europe. In addition, up to 16 DM2 patients are planned to be enrolled (sub-group - 8 active: 8 placebo).

Study drug (mexiletine 167 mg or placebo) will be started as a once a day (QD) treatment regimen. The dose will be titrated up at the Week 1 and Week 2 visits to a maximum of 1 capsule three times a day. Depending on tolerability, the dose can also be either maintained or - if required - reduced by one dose step at any time during the study to a minimum dose of 167 mg QD.

ELIGIBILITY:
Inclusion Criteria:

1. DM1 or DM2 diagnosis confirmed genetically;
2. Ability to provide informed consent;
3. Ability to understand the study requirements including intention to stay in the study until the end-of-study visit at 26 weeks of treatment;
4. Male or non-pregnant female ≥18 years of age;
5. Female patients of childbearing potential must be using an acceptable form of birth control as determined by the investigator (e.g., oral contraception, implantable, injectable/transdermal hormonal contraception, intrauterine device (IUD), barrier methods), tubal ligation, have a vasectomized partner, or are practicing abstinence;
6. No significant cardiac abnormalities as determined by a cardiologist's assessment of the electrocardiogram (ECG) and echocardiogram;
7. Capable of swallowing capsules;
8. Have sufficient finger flexor strength to grasp the handle of the dynamometer used to measure myotonia;
9. Presence of clinical handgrip myotonia (delayed relaxation of grip of ≥ 3 seconds after maximum voluntary contraction) at screening;
10. Have a Day 1 (pre-dose) handgrip dynamometer mean relaxation time of ≥1.5 seconds for the force to decline from 90% of maximum voluntary contraction force to 5%;
11. Be able to walk independently 10 meters (cane, walker, orthoses allowed);
12. DM1 patients only - Muscular impairment rating scale (MIRS) score of 2, 3, or 4.

Exclusion Criteria:

1. Are pregnant or lactating;
2. Have any one of the following medical conditions: uncontrolled diabetes mellitus, cancer other than skin cancer less than five years previously (e.g., basal-cell carcinoma (BCC) and squamous-cell carcinoma (SCC) of skin allowed), multiple sclerosis, seizure disorders, or other serious medical illness;
3. Severe renal impairment (glomerular filtration rate (GFR) < 30 mL/min);
4. Medical conditions which could interfere with muscle function such as infections, trauma, fractures, or planned surgery;
5. Medical conditions that could affect hand functioning including but not limited to rheumatoid arthritis, Dupuytren's contracture, hand deformity, etc.;
6. Severe arthritis or other medical condition (besides DM1/DM2) that would significantly impact ambulation;
7. High incidence of falls or fall-associated fractures (>5 falls during the past 12 months);
8. Preexisting elevated liver function tests > 3 times the upper limit of normal (ULN) at screening (alanine transaminase (ALT)/aspartate transaminase (AST), gamma-glutamyl transferase (GGT)) and/or any abnormal chemistry, hematology or urine lab considered clinically significant by the investigator;
9. Treatment with mexiletine within 4 weeks prior to baseline (Day 1);
10. Intake of any anti-myotonic treatment within 4 weeks prior to baseline (Day 1) such as propafenone, flecainide, lamotrigine, carbamazepine or any other channel-blocker/ anticonvulsive drugs;
11. Use of any concomitant medications that could increase the cardiac risk;
12. Known allergy to mexiletine or any local anesthetics;
13. Participation in another interventional clinical study during the last 3 months;
14. Wheelchair-bound or bed-ridden;
15. Any cardiac safety-associated condition including any of the following criteria detected by screening cardiac evaluations including 24-hour Holter monitoring, ECG, echocardiogram and clinical evaluations:

    * PR interval ≥240 ms or QRS duration ≥120 ms on resting ECG
    * Personal history of 3rd degree or 2nd degree type 2 atrioventricular block or sinus node dysfunction with pauses ≥3 seconds
    * Personal history of sustained atrial fibrillation, flutter or tachycardia (duration >30 seconds)
    * Personal history of non-sustained (ventricular triplets or more) or sustained ventricular tachycardia
    * Myocardial infarction (acute or past) or coronary artery stenosis >50%
    * New York Heart Association (NYHA) Class II to IV heart failure
    * Left ventricular systolic dysfunction with ejection fraction <50%
    * Sinus node dysfunction (including ECG sinus rate <50 beats per minute (BPM))
    * Co-administration of mexiletine and antiarrhythmics inducing torsades de pointes (class Ia: quinidine, procainamide, disopyramide, ajmaline; class Ic: encainide, flecainide, propafenone, moricizine; class III: amiodarone, sotalol, ibutilide, dofetilide, dronedarone, vernakalant)
    * Patients with implantable cardioverter defibrillators (ICDs) and pacemakers are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or non-pregnant female ≥18 years of age
Enrollment: 0 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-12 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy and safety of mexiletine for the symptomatic treatment of myotonia | 6 months
  To assess the efficacy and safety of mexiletine for the symptomatic treatment of myotonia in adult patients with myotonic dystrophy type 1 and type 2 (DM1 and DM2) by handgrip relaxation time in DM1 patients: Mean change from baseline (i.e., Day 1, pre-dose) in relaxation time of handgrip after 3 seconds of MVIC of the dominant hand using a handgrip dynamometer at Week 26. Mean relaxation time at each timepoint will be calculated from the first contraction in each of the 3 trials (each trial consists of 6 maximal voluntary contractions). Relaxation time for the assessment of myotonia will be calculated as the time required for the force to decline from 90% of maximum voluntary contraction force to 5%.

SECONDARY OUTCOMES:
To assess the efficacy of mexiletine on patient-reported outcomes by way of standardized instrument for measuring generic health status, EuroQol- 5 Dimension (EQ-5D). | Day 1 (pre-dose), Week 14, and Week 26 (or early discontinuation)
  The EQ-5D is a multi-attribute utility instrument for measuring health-related quality of life. EQ-5D: EuroQol - 5 dimensions (Health-related quality of life measure developed by EuroQol group). The index score is calculated by software hence minimum/maximum or better/worse not applicable. The EQ-5D assessments will be collected on Day 1 (pre-dose), Week 14, and Week 26 (or early discontinuation).
To assess the efficacy of mexiletine on patient-reported outcomes by Timed "Up & Go" (TUG) | 6 months
  The TUG Test (Podsiadlo, 1991; Trip 2009a) measures, in seconds, the time taken by an individual to stand up from a standard arm chair (approximate seat height of 46 cm, arm height 65 cm), walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down.
To assess the efficacy of mexiletine on patient-reported outcomes by Individualized Neuromuscular Quality of Life Questionnaire (INQoL) overall | Day 1 (pre-dose), Week 14, and Week 26 (or early discontinuation)
  INQoL- Individualized neuromuscular quality of life questionnaire. Higher score represents worsening and lower score represents better. Minimum/maximum- not applicable. The INQoL overall questionnaire will be completed on Day 1 (pre-dose), Week 14, and Week 26 (or early discontinuation)
To assess the efficacy of mexiletine on functional capacity outcome measures by Individualized Neuromuscular Quality of Life Questionnaire (INQoL) locking domain. | 6 months
  To assess the efficacy of mexiletine on functional capacity outcome measures by Individualized Neuromuscular Quality of Life Questionnaire (INQoL) locking domain.INQoL- Individualized neuromuscular quality of life questionnaire. Higher score represents worsening and lower score represents better. Minimum/maximum- not applicable.
To assess the efficacy of mexiletine on functional capacity outcome measures by Myotonia Behavior Scale (MBS). | Day 1 (pre-dose), Week 2, Week 6, Week 14, Week 18, and Week 26 (or early discontinuation)
  MBS was originally developed by Budzynski, Stoyva, Adler and Mullaney as a pain measurement instrument (Budzynski, 1973). The patient chooses one out of six framed sentences, which most closely describe the impact of the stiffness on everyday life. MBS: myotonia behavior scale, score ranges 0 - 5. Lower score is better and higher score is worsening. The MBS assessments will be completed on Day 1 (pre-dose), Week 2, Week 6, Week 14, Week 18, and Week 26 (or early discontinuation)
To assess the efficacy of mexiletine on functional capacity outcome measures by Visual Analog Scale (VAS) for myotonia. | 6 months
  The construction of VAS in this study is an absolute measure, with a straight, horizontal, 10 cm line having the endpoints "No stiffness at all" and "Stiffness as worst possible". The patient responds with a score on the line to the nearest millimeter on a 100-point scale. The VAS will be completed on Day 1 (pre-dose), Week 2, Week 6, Week 14, Week 18, and Week 26 (or early discontinuation)
To assess the efficacy of mexiletine on functional capacity outcome measures by 10 meter Walk Test (10mWT). | 6 months
  the 10mWT is a performance-based test assessing walking in two different conditions, own preferred speed and maximum speed, over a short distance. The time taken to walk 10 meters at usual comfortable and maximum speed is recorded with a stopwatch.
To assess the efficacy of mexiletine on functional capacity outcome measures by DM1-Active-c. | Day 1 (pre-dose), Week 14, and Week 26 (or early discontinuation)
  DM1-Activ-c scale is a disease-specific, Rasch-built scale, developed as a patient-reported outcome measure of capacity for activity and social participation with a 0-100 interval range (a higher score indicates higher capacity) (Hermans, 2015).VAS- Visual analogue scale. Score ranges 0-100. Lower is better and higher is worsening. The DM1-Activ-c scale score will be collected on Day 1 (pre-dose), Week 14, and Week 26 (or early discontinuation)